CLINICAL TRIAL: NCT03598803
Title: The Prevalence of Urinary Incontinence in Women and Men With Respiratory Diseases: a Questionnaire Survey
Acronym: INCONTI-SURVEY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: UIAdultsRespiratoryDisease; 2018/10JAN/006 (Other: CEHF)
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Chronic Respiratory Disease
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Urinary Incontinence Survey

SUMMARY:
Study the prevalence of the urinary incontinence among adults with respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients with chronic respiratory diseases
* Age: 18-90

Exclusion Criteria:

* Minors
* Patients with cystic fibrosis
* Cognitive disorders
* Patients who do not speak French

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with respiratory disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary Incontinence | five minutes
  Prevalence

SECONDARY OUTCOMES:
Pulmonary Function | five minutes
  VEMS

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Universitaire Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No